CLINICAL TRIAL: NCT03633669
Title: Effect of Real-world Tight Control Management of Inflammatory Bowel Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2018-07-27; First posted 2018-08-16 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tight control (Active Comparator): Group that will receive fecal calprotectin testing every 3 months
  Interventions: Diagnostic Test: Fecal calprotectin
- Standard care (Placebo Comparator): Routine clinical care
  Interventions: Other: Routine care

INTERVENTIONS:
Diagnostic Test: Fecal calprotectin — Testing every 3 months
  Arms: Tight control
Other: Routine care — As per treating gastroenterologist
  Arms: Standard care

SUMMARY:
Inflammatory bowel disease, which includes Crohn's disease and ulcerative colitis, is a condition that causes inflammation in the gastrointestinal tract. The disease goes through periods of remission and flare. Biomarkers such as fecal calprotectin have been proposed as a tool to monitor disease activity. Fecal calprotectin is a test that measures the amount of inflammation in the stool. Monitoring fecal calprotectin levels can assist gastroenterologists in making decisions regarding patients' IBD treatment such as whether to increase the dose of medications. A recent study showed that frequent measurement of fecal calprotectin every 3 months, also called the tight-control strategy, was associated with improved clinical outcomes in IBD patients. The purpose of this study is to assess whether the tight-control monitoring strategy, which includes fecal calprotectin monitoring every 3 months, improves clinical outcomes in IBD when performed in the real world compared to routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Crohn's disease or ulcerative colitis based on clinical, endoscopic, radiologic or histologic criteria.
2. Followed by a gastroenterologist at Hamilton Health Sciences, St. Joseph's Healthcare Hamilton, and London Health Sciences
3. Aged 18 or older
4. In clinical remission according to the clinical symptom assessment (Partial Mayo score < 2 or Harvey-Bradshaw Index < 4)
5. Currently treated with adalimumab

Exclusion Criteria:

1. Current abdominal abscess
2. Inability or unwillingness to provide informed consent
3. Any other condition, which in the opinion of the investigators would impede competence or compliance or possibly hinder completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Relapse | 12 months
  This will be a composite outcome of clinical symptom relapse (based on elevation of symptom scores like rise in Harvey Bradshaw Index >=3 points for Crohn's disease and Partial Mayo score >=2 points for ulcerative colitis), hospitalization, prednisone use, or IBD-related surgery

SECONDARY OUTCOMES:
Rate of Clinical symptom relapse | 12 months
  Elevation of symptom scores like rise in Harvey Bradshaw Index >= 3 points for Crohn's disease and Partial Mayo score >=2 points for ulcerative colitis
Incidence of Hospitalizations | 12 months
  Based on admission to hospital for IBD-related reasons
Incidence of change in medical therapies | 12 months
  Increased doses of current biologics, switch to different biologics, addition of immunomodulators, or steroid use would all qualify as changes in medical therapies

IPD SHARING:
Plan to Share IPD: No